CLINICAL TRIAL: NCT01341015
Title: Bedside Ultrasound in the Diagnosis of Ankle Fractures in Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0094-10
Record Dates: First submitted 2011-04-11; First posted 2011-04-25 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2011-04

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound for fracture (Experimental): All patients receive ultrasound for potential ankle fracture.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Single interventional group - patients agree to an ultrasound of potential ankle fracture, to be compared to standard of care xray.
  Other Names: ultrasound for fractures

SUMMARY:
Objectives:

A lot of children who injure their ankles come to the emergency department for an evaluation, and often an X-ray of the ankle is obtained to determine if a bone fracture is present. In more than 85% of cases, however, the injury is a sprain and not a bone fracture and can be treated with rest, ice, elevation, and pain medications. X-rays obtained in the emergency departments are time consuming, often uncomfortable for the patient, and expose children to radiation, the long-term effects of which are not yet fully understand by doctors or scientists. Bedside ultrasound is a non-invasive and a non-painful device that does not produce radiation. It was been shown to determine the presence of bone fracture in childrens' wrists and forearms just as well as X-rays do. In our study, the investigators would like to determine if a bedside ultrasound can also be used to evaluate ankle fractures in children.

Research Procedures:

In our study, the investigators will ask the parents and children, who are scheduled to get an X-ray of their ankle in the emergency department, to examine their ankles with an ultrasound machine as well. Since the bedside ultrasound is not significantly time-consuming, does not require patients to remain still, and is readily available in the department, the procedure will be performed while kids are waiting to get an X-ray, getting registered, or awaiting further treatment. On the data collection form, the investigators will document the patients' names, birthdates, medical record numbers so that their X-ray results can be compared to the ultrasound results for the purpose of the study. The information will be stored in a secure cabinet in a locked office. The investigators will also document which side is injured, where the patient feels pain and what the ankle looks like to help perform the ultrasound. The results of both the ultrasound and X-ray will be documented for each patient.

ELIGIBILITY:
Inclusion Criteria:

* age 2-18 years old
* ankle ray ordered in ER

Exclusion Criteria:

* open fracture
* multi-system trauma/other significant injuries
* history of ankle fractures? (Same ankle broken within past year)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
comparison of ultrasound to xray shows identical read | At ER visit (day 1)
  Ultrasound and the radiograph findings for each patient will be reviewed. The agreement between ultrasound and radiography will be expressed as a percentage of total number of studies performed.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Liebmann, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States